CLINICAL TRIAL: NCT03753243
Title: Phase II Study of Neoadjuvant Pembrolizumab Plus Intensive Androgen Axis Blockade Prior to Prostatectomy for High Risk Localized Prostate Cancer
Brief Title: Neoadjuvant Pembrolizumab Plus Androgen Axis Blockade Prior to Prostatectomy for High Risk Localized Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mark Garzotto, MD (U.S. Federal Agency)
Collaborators: Merck Sharp & Dohme LLC (Industry); Astellas Pharma Inc (Industry)
Responsible Party: Sponsor-Investigator, Mark Garzotto, MD, Director of Urologic Oncology, Portland VA Medical Center
Organization: Portland VA Medical Center (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15235
Record Dates: First submitted 2018-11-20; First posted 2018-11-26 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Prostate Cancer
Keywords: Neoadjuvant; Programmed cell death protein 1 (PD-1)
MeSH Terms: conditions — Prostatic Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; enzalutamide

STUDY DESIGN:
Intervention Model Description: single arm, single-stage open label Phase II of neoadjuvant immune-hormonal therapy in high-risk Localized prostate cancer.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Treatment will be planned for a total of 14 to 16 weeks. Pembrolizumab will be administered every 3 weeks via IV infusion with a dose of 200 mg per infusion. Enzalutamide will be given orally and dispensed to the patient on the date of their first infusion. The dosage of Enzalutamide will be 160 mg, administered once daily for approx. 16 weeks. GNRH agonist therapy will be administered as a standard of care therapy and will follow a standard dosage to maintain castrate levels.
  Interventions: Drug: Pembrolizumab; Drug: Enzalutamide

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg will be administered as a 30 minute IV infusion every 3 weeks.
  Other Names: Keytruda
Drug: Enzalutamide — Patients will receive daily oral doses of study drug (enzalutamide 160 mg/day), which will be administered as four capsules/day to be taken at or near the same time each day.
  Other Names: Xtandi

SUMMARY:
Pembrolizumab will be administered at a dose of 200 mg will be administered as a 30 minute IV infusion every 3 weeks. Enzalutamide will be administered at dose of 160 mg orally every day. All patients will be required to have at least one high-risk criteria.

DETAILED DESCRIPTION:
The investigators propose to study the effects of pembrolizumab combined with intensive androgen receptor (AR) targeting prior to prostatectomy with extended pelvic lymph node dissection in subjects with high-risk localized prostate cancer (HRLPC).

Trial Design- single arm, single-stage, open label Phase II of neoadjuvant immune-hormonal therapy in high-risk localized prostate cancer.

Objectives To evaluate efficacy and safety of pembrolizumab combined with intensive AR targeting prior to prostatectomy in subjects with high-risk localized prostate cancer (HRLPC).

Primary Endpoint Pathologic complete response (pCR) defined as absence of detectable malignant cells in the prostatectomy specimen evaluated by standard histologic techniques.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Capability to understand and comply with the protocol and signed informed consent document.
* Be ≥ 18 years of age on day of signing informed consent.
* Have measurable disease based on RECIST 1.1.
* Histologically confirmed, non-metastatic adenocarcinoma of the prostate
* Prostatectomy with extended lymph node dissection planned as primary therapy
* 10 year or longer life expectancy based on other co-morbidities
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Any one of the following three high risk features:

  * Gleason grade > 8-10
  * PSA > 20 ng/ml
  * Clinical stage T3a (resectable)
* No evidence of metastases .
* No other diagnosis of malignancy (with exception of non-melanoma skin cancer or a malignancy diagnosed ≥5 years ago).
* Male subjects of childbearing potential must agree to use an adequate method of contraception. Contraception, starting with the first dose of study therapy through the time of surgery. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Demonstrate adequate organ function, all screening labs should be performed within 30 days of treatment initiation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2018-12-03 (Actual); Primary Completion 2022-09-03 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response | 4 months
  No cancer detected on pathology examination of prostatectomy specimen

SECONDARY OUTCOMES:
Treatment Related Adverse Events | 4 months + 30 days
  Grade 3 or higher adverse event (AE) possibly related or related to any of three treatment drugs (pembrolizumab, enzalutamide, Gonadotropin-releasing hormone (GNRH) agonist) per CTCAE v4.03, evaluated up until 30 days after prostatectomy
Immune -related Adverse Events | 4 months + 30 days
  Grade 2 or higher immune related AE possibly related or related to any of three treatment drugs (pembrolizumab, enzalutamide, GNRH agonist) per CTCAE v4.03, evaluated up until 30 days after prostatectomy
Biochemical Complete Response | 4 months
  Prostate-Specific Antigen (PSA) < 0.1 ng/mL prior to prostatectomy
Incidence of Surgical Complications | 4 months
  Clavien-Dindo Classification of Surgical Complications compared to historical department incidence rates.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Garzotto, MD, Principal Investigator — Portland VA Medical Center
Locations (1):
- VA Portland Healthcare System, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pala L, De Pas T, Conforti F. Boosting anticancer immunotherapy through androgen receptor blockade. Cancer Cell. 2022 May 9;40(5):455-457. doi: 10.1016/j.ccell.2022.04.007. Epub 2022 May 9. PMID 35537411

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-13): https://cdn.clinicaltrials.gov/large-docs/43/NCT03753243/Prot_SAP_000.pdf